CLINICAL TRIAL: NCT07340632
Title: BLOOM43 for Preconditioning (B4P): A Pilot Study to Evaluate the Use of the Plexaa Preconditioning Device (BLOOM43) for Reconstructive Breast Surgery - A Prospective Cohort Multicentre Study
Brief Title: B4P Trial - BLOOM43 for Preconditioning
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Plexaa Ltd (Industry)
Collaborators: Royal Marsden NHS Foundation Trust (Other); Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B4PTrial; NIHR206435 (Other: National Institute for Health and Care Research (NIHR))
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Skin Necrosis; Breast Reconstruction; Breast Surgery
Keywords: Mastectomy skin flap necrosis; Breast reconstruction; Breast surgery; Preconditioning; Skin necrosis
MeSH Terms: conditions — Necrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (single arm) (Experimental): Each patient will be given the device, BLOOM43, for use at home. It will be worn in a patient's existing bra over their ipsilateral breast (the breast to be operated on) and the preconditioning protocol will be undertaken 12 hours before surgery - i.e. the evening before. Patients will then attend hospital for their breast surgery the next day as planned. For the patients undergoing bilateral skin/nipple-sparing mastectomy with immediate reconstruction, they will be asked to precondition only the right breast.
  Interventions: Device: BLOOM43

INTERVENTIONS:
Device: BLOOM43 — BLOOM43 works by delivering heat preconditioning to the breast skin before surgery.

SUMMARY:
The goal of this clinical trial is to evaluate the use of the Plexaa preconditioning device (BLOOM43) in patients undergoing reconstructive breast surgery for breast cancer. This study aims to understand a participant's experience of the device, including its usability and acceptability.

Participants will use the device to precondition their breast the evening before undergoing surgery (mastectomy with immediate autologous and/or implant-based reconstruction).

ELIGIBILITY:
Inclusion Criteria:

* All females over the age of 18 years (no maximum age limit)
* Patients undergoing skin-sparing mastectomy or nipple-sparing mastectomy and immediate breast reconstruction (autologous and/or implant)

Exclusion Criteria:

* Delayed (two-stage) breast reconstruction patients
* Patients undergoing simple mastectomy or wide local excision of a breast tumour
* Inflammatory breast cancer patients
* Presence of open breast skin wounds, or infected or inflamed breast skin
* Presence of a cardiac pacemaker, defibrillator or any other implantable electronic device

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-16 (Estimated); Primary Completion 2026-09-16 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Participant experience | 30 days
  Participants' experience of the device will be evaluated with the use of a questionnaire. Most of the questions will consist of multiple-choice components with a five-point scale and there will also be a section for further comments from participants.

SECONDARY OUTCOMES:
Mastectomy skin flap necrosis | 90 days
  Proportion of participants experiencing mastectomy skin flap necrosis and the rates of hospital re-admission and surgical re-intervention due to this
Compliance | 1 day
  Proportion of participants who are compliant with the preconditioning protocol

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeevan R, Cromwell DA, Browne JP, Caddy CM, Pereira J, Sheppard C, Greenaway K, van der Meulen JH. Findings of a national comparative audit of mastectomy and breast reconstruction surgery in England. J Plast Reconstr Aesthet Surg. 2014 Oct;67(10):1333-44. doi: 10.1016/j.bjps.2014.04.022. Epub 2014 May 14. PMID 24908545
- [Background] Robertson SA, Jeevaratnam JA, Agrawal A, Cutress RI. Mastectomy skin flap necrosis: challenges and solutions. Breast Cancer (Dove Med Press). 2017 Mar 13;9:141-152. doi: 10.2147/BCTT.S81712. eCollection 2017. PMID 28331365
- [Background] Mehta S, Rolph R, Cornelius V, Harder Y, Farhadi J. Local heat preconditioning in skin sparing mastectomy: a pilot study. J Plast Reconstr Aesthet Surg. 2013 Dec;66(12):1676-82. doi: 10.1016/j.bjps.2013.07.034. Epub 2013 Sep 4. PMID 24011908
- [Background] Kankam HKN, Mehta S, Jain A. Thermal Preconditioning for Surgery: A Systematic Review. J Plast Reconstr Aesthet Surg. 2020 Sep;73(9):1645-1664. doi: 10.1016/j.bjps.2020.05.025. Epub 2020 May 21. PMID 32505626
- [Background] Mehta S, Cro SC, Coomber B, Rolph R, Cornelius V, Farhadi J. A randomised controlled feasibility trial to evaluate local heat preconditioning on wound healing after reconstructive breast surgery: the preHEAT trial. Pilot Feasibility Stud. 2019 Jan 11;5:5. doi: 10.1186/s40814-019-0392-y. eCollection 2019. PMID 30656059